CLINICAL TRIAL: NCT00184171
Title: Treatment of Microscopic Colitis (Collagenous Colitis and Lymphocytic Colitis) With Budesonide, Bismuth or Fiber
Brief Title: Treatment of Microscopic Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient data quality
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLV 01-07035
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Colitis
Keywords: Microscopic colitis; Drug treatment; Diarrhoea
MeSH Terms: conditions — Colitis; Colitis, Microscopic; Diarrhea | interventions — Budesonide; Bismuth; Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Budesonide (Experimental): Budesonide 9mg
  Interventions: Drug: Budesonide
- bismuth (Experimental): Bismuth mixture
  Interventions: Drug: Bismuth
- Fiber (Sham Comparator): Fiber preparation
  Interventions: Drug: Fiber

INTERVENTIONS:
Drug: Budesonide — Budesonide 9 mg
  Arms: Budesonide
Drug: Bismuth — Bismuth mixture
  Arms: bismuth
Drug: Fiber — Fiber for control
  Arms: Fiber

SUMMARY:
The study compares the effect of Budesonide, Bismuth and fiber in patients with microscopic colitis

DETAILED DESCRIPTION:
This randomized, controlled, open study compares the effects of 8 weeks' treatment with Budesonide, Bismuth and fiber on symptoms and histological findings in patients with microscopic colitis (both collagenous colitis and lymphocytic colitis).

ELIGIBILITY:
Inclusion Criteria:

* Microscopic colitis verified with biopsies from the colon
* Symptoms to such an extent that treatment is indicated
* Age > 17 years
* Informed consent

Exclusion Criteria:

* Previous treatment with any of the investigational drugs
* Patients treated with ketoconazole
* Pregnant and breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-11; Primary Completion 2010-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Symptoms: Stool frequency and consistency | 2001 - 2011
  September 2010: Patient's enrollment completed. Data analysis ongoing.

SECONDARY OUTCOMES:
Histological findings in biopsies from colon | 2001 - 2011
  Patient's enrollment completed. Data analysis ongoing.

CONTACTS AND LOCATIONS:
Overall Officials: Per G Farup, PhD, Study Chair — Norwegian University of Science and Technology
Locations (9):
- Norway (9):
  - Aust-Agder Sentralsjukehus, Arendal
  - Sykehuset Innlandet HF, Gjøvik, Gjøvik
  - Sykehuset Innlandet, HF, Hamar, Hamar
  - Sykehuset Innlandet HF, Lillehammer, Lillehammer
  - Helse NordMøre og Romsdal, Molde
  - Akershus Universitetssykehus, Nordbyhagen
  - Aker sykehus, Oslo
  - Rikshopitalet, Oslo
  - St. Olavs Hospital, Trondheim